CLINICAL TRIAL: NCT00138554
Title: Extension to a Study on the Efficacy and Safety of Vildagliptin in Combination With Pioglitazone in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLAF237A2304E1
Record Dates: First submitted 2005-08-27; First posted 2005-08-30 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- vildagliptin 50 mg qd + pioglitazone 45 mg qd (Experimental): vildagliptin 50 mg qd + pioglitazone 45 mg qd for 28 weeks
  Interventions: Drug: vildagliptin; Drug: pioglitazone
- vildagliptin 50 mg bd+ pioglitazone 45 mg qd (Experimental): vildagliptin 50 mg bd + pioglitazone 45 mg qd for 28 weeks
  Interventions: Drug: vildagliptin; Drug: pioglitazone

INTERVENTIONS:
Drug: vildagliptin
Drug: pioglitazone — pioglitazone 45 mg qd

SUMMARY:
Many people with type 2 diabetes cannot maintain target blood glucose levels when taking a single oral drug. This is a 28-week extension to a study to assess the safety and effectiveness of vildagliptin, an unapproved drug, in lowering overall blood glucose levels when added to pioglitazone in people with type 2 diabetes not at target blood glucose levels on pioglitazone or rosiglitazone alone. The purpose of the extension study is to gather data on the long-term safety and effectiveness of vildagliptin in people with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Only patients successfully completing study CLAF237A2304 are eligible
* Written informed consent
* Ability to comply with all study requirements

Exclusion Criteria:

* Premature discontinuation from study CLAF237A2304
* Other protocol-defined exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2004-11; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Safety of vildagliptin in combination with pioglitazone during 52 weeks of treatment
Change from baseline in HbA1c at 52 weeks

SECONDARY OUTCOMES:
Change in HbA1c between 24 weeks and 52 weeks
Change from baseline in fasting plasma glucose at 52 weeks
Change in fasting plasma glucose between 24 weeks and 52 weeks
Change from baseline in HOMA B at 52 weeks
Change from baseline in HOMA IR at 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States

REFERENCES:
- [Result] Ligueros-Saylan M, Foley JE, Schweizer A, Couturier A, Kothny W. An assessment of adverse effects of vildagliptin versus comparators on the liver, the pancreas, the immune system, the skin and in patients with impaired renal function from a large pooled database of Phase II and III clinical trials. Diabetes Obes Metab. 2010 Jun;12(6):495-509. doi: 10.1111/j.1463-1326.2010.01214.x. PMID 20518805